CLINICAL TRIAL: NCT04729621
Title: A Randomized, Double-Blind, Multinational, Multicenter Study to Compare Efficacy, Safety, and Immunogenicity of TVB-009P and Denosumab (Prolia®) in Patients With Postmenopausal Osteoporosis
Brief Title: A Study to Test if TVB-009P is Effective in Relieving Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TVB009-IMB-30085
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- TVB-009 main treatment period (Experimental): TVB-009 (denosumab) pre-filled syringe, administered at weeks 1 and 26
  Interventions: Combination Product: TVB-009
- PROLIA main treatment period (Active Comparator): Prolia® (denosumab) pre-filled syringe, administered at weeks 1 and 26
  Interventions: Combination Product: Prolia®
- TVB-009 main / TVB-009 transition period (Experimental): TVB-009 (denosumab) pre-filled syringe, administered at week 52 in patients that were randomized to TVB-009 in the main treatment period
  Interventions: Combination Product: TVB-009
- PROLIA main / PROLIA transition period (Active Comparator): Prolia® (denosumab) pre-filled syringe, administered at week 52 in patients that were randomized to PROLIA in the main treatment period
  Interventions: Combination Product: Prolia®
- PROLIA main / TVB-009 transition period (Experimental): TVB-009 (denosumab) pre-filled syringe, administered at week 52 in patients that were randomized to PROLIA in the main treatment period
  Interventions: Combination Product: TVB-009; Combination Product: Prolia®

INTERVENTIONS:
Combination Product: TVB-009 — TVB-009 Denosumab solution for injection 60 mg/mL (1 mL) prefilled syringe (PFS)
  Arms: PROLIA main / TVB-009 transition period; TVB-009 main / TVB-009 transition period; TVB-009 main treatment period
Combination Product: Prolia® — Denosumab solution for injection 60 mg/mL (1 mL) prefilled syringe (PFS)
  Arms: PROLIA main / PROLIA transition period; PROLIA main / TVB-009 transition period; PROLIA main treatment period

SUMMARY:
The purpose of this study is to demonstrate similar efficacy and safety between TVB-009 and Prolia® (denosumab)

DETAILED DESCRIPTION:
This is a multinational, multicenter, randomized, double-blind study to demonstrate similar efficacy and safety of TVB-009 compared to Prolia® administered subcutaneously at doses of 60 mg every 26 weeks. Approximately 326 postmenopausal women with osteoporosis will be randomized to receive either TVB-009 or Prolia®. At week 52, patients in the Prolia® arm will be re-randomized 1:1 to either continue with a third dose of Prolia® or transition to TVB-009 and receive a single dose of TVB-009 in the transition period to assess immunogenicity and safety after a transition from Prolia® to TVB-009. The total treatment duration for each patient is 78 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal womeen (≥60 and ≤90 years) with a diagnosis of osteoporosis
* Body weight ≥50 kg and ≤90 kg
* Bone Mineral Density (BMD) measurement T score of less than -2.5 but not less than -4.0 by dual-energy X-ray absorptiometry (DXA) at the lumbar spine at screening
* At least 3 vertebrae in the L1 L4 region that are evaluable by dual-energy X-ray absorptiometry (DXA)

Exclusion Criteria:

* One severe or more than two moderate vertebral fractures
* History and/or presence of hip fracture or atypical femur fracture
* Any prior treatment with denosumab
* Ongoing use of any bone active drugs which can affect Bone Mineral Density (BMD)
* Vitamin D deficiency or hyper- or hypocalcemiacium at screening
* Hyperthyroidism, hypothyroidism, hypoparathyroidism or hyperparathyroidism
* Any medical condition that could jeopardize or would compromise the patient's safety or ability to participate in this study

Other Inclusion/exclusion criteria may apply

Ages: 60 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Pharmaceuticals, Inc.
Locations (78):
- United States (20):
  - Teva Site 103, Phoenix, Arizona
  - Teva Site 119, Tucson, Arizona
  - Teva Site 118, San Diego, California
  - Teva Site 107, New London, Connecticut
  - Teva Site 115, Coral Gables, Florida
  - Teva Site 114, Edgewater, Florida
  - Teva Site 116, Lake City, Florida
  - Teva Site 109, Miami Lakes, Florida
  - Teva Site 117, Miami Springs, Florida
  - Teva Site 110, Oldsmar, Florida
  - Teva Site 120, Orlando, Florida
  - Teva Site 102, Ormond Beach, Florida
  - Teva Site 101, Port Saint Lucie, Florida
  - Teva Site 111, Sarasota, Florida
  - Teva Site 104, Tamarac, Florida
  - Teva Site 112, Henderson, Nevada
  - Teva Site 113, North Las Vegas, Nevada
  - Teva Site 105, Albuquerque, New Mexico
  - Teva Site 108, Duncansville, Pennsylvania
  - Teva Site 106, Seattle, Washington
- Bulgaria (10):
  - Teva Site 203, Blagoevgrad
  - Teva Site 207, Dimitrovgrad
  - Teva Site 252, Haskovo
  - Teva Site 202, Lom
  - Teva Site 205, Plovdiv
  - Teva Site 250, Silistra
  - Teva Site 201, Sofia
  - Teva Site 204, Sofia
  - Teva Site 251, Sofia
  - Teva Site 206, Stara Zagora
- Czechia (6):
  - Teva Site 211, Brno
  - Teva Site 213, Ostrava
  - Teva Site 212, Pardubice
  - Teva Site 209, Prague
  - Teva Site 210, Prague
  - Teva Site 208, Uherské Hradiště
- Georgia (6):
  - Teva Site 214, Tbilisi
  - Teva Site 215, Tbilisi
  - Teva Site 216, Tbilisi
  - Teva Site 217, Tbilisi
  - Teva Site 218, Tbilisi
  - Teva Site 219, Tbilisi
- Germany (4):
  - Teva Site 223, Dresden
  - Teva Site 220, Hamburg
  - Teva Site 221, Nümbrecht
  - Teva Site 222, Würzburg
- Hungary (5):
  - Teva Site 226, Balatonfüred
  - Teva Site 225, Budapest
  - Teva Site 227, Budapest
  - Teva Site 253, Budapest
  - Teva Site 224, Nyíregyháza
- Poland (6):
  - Teva Site 228, Bialystok
  - Teva Site 233, Krakow
  - Teva Site 231, Lodz
  - Teva Site 230, Warsaw
  - Teva Site 232, Warsaw
  - Teva Site 229, Wroclaw
- Russia (8):
  - Teva Site 235, Moscow
  - Teva Site 236, Saint Petersburg
  - Teva Site 254, Saint Petersburg
  - Teva Site 255, Saint Petersburg
  - Teva Site 256, Saint Petersburg
  - Teva Site 257, Saint Petersburg
  - Teva Site 234, Yaroslavl
  - Teva Site 258, Yaroslavl
- Slovakia (6):
  - Teva Site 238, Bratislava
  - Teva Site 242, Bratislava
  - Teva Site 237, Hlohovec
  - Teva Site 241, Lučenec
  - Teva Site 240, Ľubochňa
  - Teva Site 239, Prešov
- Ukraine (7):
  - Teva Site 244, Kyiv
  - Teva Site 245, Kyiv
  - Teva Site 247, Kyiv
  - Teva Site 248, Kyiv
  - Teva Site 249, Kyiv
  - Teva Site 243, Vinnytsia
  - Teva Site 246, Zaporizhia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 332 subjects were randomized into the study. Those that completed the Main treatment period were then randomized into the transition period. Therefore, the 3 arms noted as "Transition period" are the same subjects that were included in the "Treatment Period".
Period: Main Treatment Period (Week1 to Week 52)
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period | TVB-009 Main / TVB-009 Transition Period | PROLIA Main / PROLIA Transition Period | PROLIA Main / TVB-009 Transition Period
Started | 166 | 166 | 0 | 0 | 0
Completed | 148 | 143 | 0 | 0 | 0
Not Completed | 18 | 23 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 7 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 13 | 12 | 0 | 0 | 0
Not completed — Multiple Other Reasons | 2 | 4 | 0 | 0 | 0
Period: Transition Period (Week 52 to Week 78)
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period | TVB-009 Main / TVB-009 Transition Period | PROLIA Main / PROLIA Transition Period | PROLIA Main / TVB-009 Transition Period
Started (Subjects who completed the Main Treatment Period were re-randomized to one of 3 new arms.) | 0 | 0 | 148 | 72 | 71
Completed | 0 | 0 | 140 | 67 | 69
Not Completed | 0 | 0 | 8 | 5 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 7 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Multiple Other Reasons | 0 | 0 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The baseline characteristics are only presented for the Treatment Period Arms as the same subject were employed in the Transition Period.
Groups:
- Total: Total of all reporting groups
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period | Total
Number analyzed (Participants) | 166 | 166 | 332
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (5.69) | 67.7 (5.56) | 68.1 (5.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166 | 166 | 332
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 18 | 41
  Not Hispanic or Latino | 143 | 148 | 291
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 165 | 164 | 329
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Hungary | 11 | 6 | 17
  United States | 34 | 35 | 69
  Czechia | 21 | 19 | 40
  Ukraine | 13 | 12 | 25
  Poland | 30 | 37 | 67
  Georgia | 17 | 9 | 26
  Slovakia | 6 | 13 | 19
  Bulgaria | 22 | 20 | 42
  Germany | 1 | 1 | 2
  Russia | 11 | 14 | 25
Previous Use of Biophosphonates [Count of Participants; unit: Participants]
  Yes | 21 | 21 | 42
  No | 145 | 145 | 290
Prior Fractures [Count of Participants; unit: Participants]
  Yes | 37 | 38 | 75
  No | 129 | 128 | 257
Taking Calcium & Vitamin D Supplements [Count of Participants; unit: Participants] — Population: Calcium & Vitamin D Supplement status was only required for patients that experienced any fractures prior to study start.
  Participants
    number analyzed (Participants) | 37 | 38 | 75
    Yes | 28 | 28 | 56
    No | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LS-BMD at Week 52
Description: Percent change from baseline in lumbar spine bone mineral density (LS BMD) based on centrally assessed dual energy X ray absorptiometry (DXA) at week 52
Time Frame: Baseline and week 52
Population: The mITT population was used for this analysis. The modified intent-to-treat (mITT) analysis set will include all randomized patients who received at least 1 dose of IMP and had at least 1 post-baseline evaluation of LS-BMD
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change from baseline
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period
Number analyzed (Participants) | 157 | 152
percentage of change from baseline | 4.76 [3.82 to 5.69] | 4.54 [3.62 to 5.47]
Statistical Analysis 1: Comparison: TVB-009 Main Treatment Period vs PROLIA Main Treatment Period; LS means, differences and confidence intervals (CI) from the ANCOVA model with percent change from baseline to Week 52 in LS-BMD as the outcome, treatment group, region and previous use of bisphosphates as fixed effects, baseline LS-BMD and baseline weight as covariates. Missing outcomes imputed using multiple imputation methods under the MAR assumption; Test type: Equivalence — Biosimilarity will be demonstrated if the 95% CI for the difference falls entirely within the equivalence margin of (-1.45, +1.45); Mean Difference (Net) = 0.21, 95% CI 2-sided [-0.73 to 1.15]

2. Secondary Outcome: Percent Change From Baseline in sCTX-1 at Week 26
Description: Percent change from baseline in serum C-telopeptide cross-link of type 1 collagen at week 26
Time Frame: Baseline and week 26
Population: The mITT was used for this analysis. The modified intent-to-treat (mITT) analysis set includes all randomized patients who received at least 1 dose of IMP and had at least 1 post-baseline evaluation of LS-BMD
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change from baseline
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period
Number analyzed (Participants) | 157 | 152
percentage of change from baseline | -56.05 [-64.99 to -47.12] | -65.13 [-74.09 to -56.17]
Statistical Analysis 1: Comparison: TVB-009 Main Treatment Period vs PROLIA Main Treatment Period; LS means, differences and confidence intervals (CI) from the ANCOVA model with percent change from baseline to Week 26 in sCTX-1 as the outcome, treatment group, region and previous use of bisphosphates as fixed effects, baseline sCTX-1 and baseline weight as covariates. Missing outcomes are not imputed. Results below the limit of quantification (BLQ) are imputed as the low limit of quantification (LLOQ = 0.033 ng/mL); Test type: Equivalence — Biosimilarity will be demonstrated if the 95% CI for the difference falls entirely within the equivalence margin of (-20, +20); Mean Difference (Net) = 9.07, 95% CI 2-sided [-0.14 to 18.29]

3. Secondary Outcome: Percent Change From Baseline in LS-BMD at Week 26
Description: Percent change from baseline in lumbar spine bone mineral density (LS BMD) based on centrally assessed dual energy X ray absorptiometry (DXA) at week 26
Time Frame: Baseline and week 26
Population: The mITT population was used in this analysis.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period
Number analyzed (Participants) | 157 | 151
percentage of change from baseline | 3.70 (4.294) | 3.62 (3.815)

4. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD at Week 26
Description: Percent change from baseline in femoral neck bone mineral density (BMD) based on centrally assessed dual energy X ray absorptiometry (DXA)at week 26
Time Frame: Baseline, week 26
Population: mITT population was used for this analysis.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period
Number analyzed (Participants) | 156 | 150
percentage of change from baseline | 1.87 (4.877) | 2.01 (3.611)

5. Secondary Outcome: Percent Change From Baseline in Total Hip BMD at Week 26
Description: Percent change from baseline in total hip bone mineral density (BMD) based on centrally assessed dual energy X ray absorptiometry (DXA) at week 26
Time Frame: Baseline, week 26
Population: mITT population was used for the analysis.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period
Number analyzed (Participants) | 156 | 150
percentage of change from baseline | 1.89 (3.488) | 2.02 (2.526)

6. Secondary Outcome: Percent Change From Baseline in sCTX-1
Description: Percent change from baseline in serum C-telopeptide cross-link of type 1 collagen
Time Frame: Baseline through Week 52
Population: mITT population was used for this analysis.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period
Number analyzed (Participants) | 151 | 146
percentage of change from baseline | -57.91 (44.161) | -68.80 (35.846)

7. Secondary Outcome: Percentage of Participatns With sCTX-1 Suppression at Week 4
Description: Proportion of patients with suppression of serum C-telopeptide cross-link of type 1 collagen at week 4
Time Frame: Week 4
Population: mITT population was used.
Measure: Number; unit: Percentage of participants
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period
Number analyzed (Participants) | 155 | 151
Percentage of participants | 94.2 | 94.0

8. Secondary Outcome: Percent Change From Baseline in P1NP
Description: Percent change from baseline in procollagen type 1 N propeptide (P1NP) to Week 52
Time Frame: Baseline through Week 52
Population: mITT population was used for this analysis.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period
Number analyzed (Participants) | 151 | 146
percentage of change from baseline | -56.43 (35.431) | -62.03 (33.712)

9. Secondary Outcome: Number of Fractures up to Week 52
Description: Number of patients with who experienced any new fractures up to week 52.
Time Frame: Up to week 52
Population: mITT population was used.
Measure: Number; unit: number participants with fractures
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period
Number analyzed (Participants) | 157 | 152
number participants with fractures | 3 | 5

10. Secondary Outcome: Percent Change From Week 52 in LS-BMD by DXA at Week 78
Description: Percent change from week 52 in lumbar spine bone mineral density (LS BMD) based on centrally assessed dual energy X ray absorptiometry (DXA) at week 78
Time Frame: Week 52 through week 78
Population: TmITT population was used. The transition modified intent-to-treat (TmITT) analysis set will include all patients who received the third dose of IMP and had an end-of-study evaluation of LS-BMD.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | TVB-009 Main / TVB-009 Transition Period | PROLIA Main / PROLIA Transition Period | PROLIA Main / TVB-009 Transition Period
Number analyzed (Participants) | 137 | 62 | 68
percentage of change from baseline | 0.82 (3.120) | 1.15 (3.440) | 1.24 (3.069)

11. Secondary Outcome: Percent Change From Week 52 in Femoral Neck BMD by DXA at Week 78
Description: Percent change from week 52 in femoral neck bone mineral density (LS BMD) based on centrally assessed dual energy X ray absorptiometry (DXA) at week 78
Time Frame: Week 52 through week 78
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percent change from week 52
Arm/Group | TVB-009 Main / TVB-009 Transition Period | PROLIA Main / PROLIA Transition Period | PROLIA Main / TVB-009 Transition Period
Number analyzed (Participants) | 137 | 62 | 68
Percent change from week 52 | 0.38 (3.525) | 0.80 (3.560) | 0.94 (3.082)

12. Secondary Outcome: Percent Change From Week 52 in Total Hip BMD by DXA at Week 78
Description: Percent change from week 52 in total hip bone mineral density (LS BMD) based on centrally assessed dual energy X ray absorptiometry (DXA) at week 78
Time Frame: Week 52 through week 78
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percent change from week 52
Arm/Group | TVB-009 Main / TVB-009 Transition Period | PROLIA Main / PROLIA Transition Period | PROLIA Main / TVB-009 Transition Period
Number analyzed (Participants) | 137 | 62 | 68
Percent change from week 52 | 0.01 (2.089) | 0.66 (2.109) | 0.27 (2.264)

13. Secondary Outcome: Difference Between Percent Change From Baseline in sCTX-1 Between Week 52 and Week 78
Description: Difference in the percent change from baseline in serum C-telopeptide cross-link of type 1 collagen from baseline to Week 78 as compared to baseline to Week 52
Time Frame: Baseline, Week 52, Week 78
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | TVB-009 Main / TVB-009 Transition Period | PROLIA Main / PROLIA Transition Period | PROLIA Main / TVB-009 Transition Period
Number analyzed (Participants) | 137 | 63 | 69
Percent change from baseline | 9.95 (41.612) | 13.17 (28.558) | 7.55 (36.509)

14. Secondary Outcome: Difference Between Percent Change From Baseline in P1NP Between Week 52 and Week 78
Description: The difference in the Percent change from baseline in procollagen type 1 N propeptide at Week 78 compared to Week 52.
Time Frame: Baseline, Week 52, Week 78
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | TVB-009 Main / TVB-009 Transition Period | PROLIA Main / PROLIA Transition Period | PROLIA Main / TVB-009 Transition Period
Number analyzed (Participants) | 137 | 63 | 69
Percent change | 3.95 (23.376) | 4.83 (14.551) | 2.89 (39.804)

15. Secondary Outcome: Number of Patients With Fractures Between Week 52 and Week 78
Description: Number of patients experiencing new fractures between week 52 and week 78
Time Frame: Week 52 through week 78
Population: as for outcome 10
Measure: Number; unit: Number participants with fractures
Arm/Group | TVB-009 Main / TVB-009 Transition Period | PROLIA Main / PROLIA Transition Period | PROLIA Main / TVB-009 Transition Period
Number analyzed (Participants) | 138 | 64 | 69
Number participants with fractures | 1 | 0 | 1

16. Secondary Outcome: Incidence of Adverse Event
Description: Number of patients reporting at least one treatment-emergent adverse event up to week 52
Time Frame: Up to week 52
Population: Safety Analysis Set (SAS) was used. The safety analysis set will include all randomized patients who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period
Number analyzed (Participants) | 166 | 165
Participants
  TEAE Related to Study Drug | 19 | 13
  TEAE Related to Medical Device | 0 | 0
  TEAE Not Related to Study Drug | 104 | 95
  No TEAEs Reported | 43 | 57

17. Secondary Outcome: Incidence of Adverse Events in the Transition Period
Description: Number of patients reporting at least one treatment-emergent adverse event between weeks 52 and 78
Time Frame: Week 52 through week 78
Population: Transition Safety Analysis Set was used. The transition safety analysis set will include all patients who received the third dose of the IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | TVB-009 Main / TVB-009 Transition Period | PROLIA Main / PROLIA Transition Period | PROLIA Main / TVB-009 Transition Period
Number analyzed (Participants) | 148 | 72 | 71
Participants
  TEAE Related to Study Drug | 2 | 0 | 0
  TEAE Related to Medical Device | 0 | 0 | 0
  TEAE Not Related to Study Drug | 48 | 20 | 26
  No TEAE Reported | 98 | 52 | 45

18. Secondary Outcome: Incidence of Antidrug Antibodies (ADAs) in the Main Treatment Period
Description: Number of patients with confirmed positive antidrug antibodies (ADAs) post-baseline through Week 52
Time Frame: Anytime Post Baseline through Week 52
Population: The Safety Analysis Set was used. The safety analysis set will include all randomized patients who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period
Number analyzed (Participants) | 166 | 165
Participants
  ADA Status: Positive | 11 | 25
  ADA Status: Positive, Not Treatment Related | 8 | 11
  ADA Status: Negative | 147 | 129
  Neutralizing ADA Status Among Positive: number analyzed (Participants) | 11 | 25
  Neutralizing ADA Status Among Positive: Positive | 1 | 2
  Neutralizing ADA Status Among Positive: Positive, Not Treatment Related | 0 | 0
  Neutralizing ADA Status Among Positive: Negative | 10 | 23

19. Secondary Outcome: Incidence of Antidrug Antibodies (ADAs) in the Transition Period
Description: Number of patients with confirmed positive antidrug antibodies (ADAs) at Week 65
Time Frame: Anytime in Week 52 through Week 78
Population: The Transition Safety Analysis Set was used. The transition safety analysis set will include all patients who received the third dose of the IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | TVB-009 Main / TVB-009 Transition Period | PROLIA Main / PROLIA Transition Period | PROLIA Main / TVB-009 Transition Period
Number analyzed (Participants) | 147 | 70 | 70
Participants
  ADA Status: Positive | 7 | 5 | 4
  ADA Status: Positive, Not Treatment Related | 7 | 4 | 1
  ADA Status: Negative | 133 | 61 | 65
  Neutralizing ADA Status Among Positive: number analyzed (Participants) | 7 | 5 | 4
  Neutralizing ADA Status Among Positive: Positive | 1 | 0 | 0
  Neutralizing ADA Status Among Positive: Positive, Not Treatment Related | 0 | 0 | 0
  Neutralizing ADA Status Among Positive: Negative | 6 | 5 | 4

20. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD at Week 52
Description: Percent change from baseline in femoral neck bone mineral density (BMD) based on centrally assessed dual energy X ray absorptiometry (DXA)at week 52
Time Frame: Baseline through Week 52
Population: mITT population was used for this analysis.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period
Number analyzed (Participants) | 150 | 145
Percent change from baseline | 2.39 (5.795) | 2.34 (3.780)

21. Secondary Outcome: Percent Change From Baseline in Total Hip BMD at Week 52
Description: Percent change from baseline in total hip bone mineral density (BMD) based on centrally assessed dual energy X ray absorptiometry (DXA) at week 52
Time Frame: Baseline through Week 52
Population: mITT population was used for the analysis.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period
Number analyzed (Participants) | 150 | 145
Percent change from baseline | 2.67 (3.981) | 3.00 (2.768)

22. Secondary Outcome: Number of TEAEs Leading to Patient Withdraw From the Study
Description: Number of patients that withdraw or are removed from the study due to treatment emergent adverse events from both the main and transition treatment periods.
Time Frame: Main Treatment Period = Baseline-Week 52; Transition period = Week 52-78
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period | TVB-009 Main / TVB-009 Transition Period | PROLIA Main / PROLIA Transition Period | PROLIA Main / TVB-009 Transition Period
Number analyzed (Participants) | 166 | 165 | 148 | 72 | 71
Participants | 3 | 7 | 0 | 0 | 0

23. Secondary Outcome: Local Tolerability at Injection Site
Description: Number of patients who report Injection Site Reactions at Day 1, Week 26, or Week 52.
Time Frame: Main Treatment Period = Day 1 & Week 26; Transition Treatment Period = Week 52
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period | TVB-009 Main / TVB-009 Transition Period | PROLIA Main / PROLIA Transition Period | PROLIA Main / TVB-009 Transition Period
Number analyzed (Participants) | 166 | 165 | 148 | 72 | 71
Participants
  Day 1: number analyzed (Participants) | 166 | 165 | 0 | 0 | 0
  Day 1: Erythema | 5 | 4 |  |  |
  Day 1: Ecchymosis | 4 | 2 |  |  |
  Day 1: Induration | 2 | 3 |  |  |
  Day 1: Tenderness | 3 | 4 |  |  |
  Day 1: Warmth | 0 | 1 |  |  |
  Day 1: Swelling | 2 | 1 |  |  |
  Day 1: Pain | 6 | 5 |  |  |
  Day 1: No Reaction | 144 | 145 |  |  |
  Week 26: number analyzed (Participants) | 158 | 153 | 0 | 0 | 0
  Week 26: Erythema | 2 | 4 |  |  |
  Week 26: Ecchymosis | 3 | 0 |  |  |
  Week 26: Induration | 2 | 0 |  |  |
  Week 26: Tenderness | 1 | 1 |  |  |
  Week 26: Warmth | 0 | 1 |  |  |
  Week 26: Swelling | 1 | 1 |  |  |
  Week 26: Pain | 7 | 4 |  |  |
  Week 26: No Reaction | 142 | 142 |  |  |
  Week 52: number analyzed (Participants) | 0 | 0 | 148 | 72 | 71
  Week 52: Erythema |  |  | 2 | 2 | 2
  Week 52: Ecchymosis |  |  | 3 | 0 | 1
  Week 52: Induration |  |  | 3 | 3 | 0
  Week 52: Tenderness |  |  | 1 | 1 | 1
  Week 52: Warmth |  |  | 0 | 2 | 0
  Week 52: Swelling |  |  | 0 | 1 | 1
  Week 52: Pain |  |  | 6 | 4 | 3
  Week 52: No Reaction |  |  | 133 | 59 | 63

ADVERSE EVENTS:
Time Frame: The Main Treatment Period collected adverse event data for a 52 week period (baseline to week 52). The transitional period collected adverse event data for a 26 week period (week 52 to week 78).
Description: All adverse events were coded using the Medical Dictionary for Regulatory Activities (MedDRA). Each patient will be counted only once in each preferred term (PT) or system organ class (SOC) category for the analyses of safety.
Arm/Group | TVB-009 Main Treatment Period | PROLIA Main Treatment Period | TVB-009 Main / TVB-009 Transition Period | PROLIA Main / PROLIA Transition Period | PROLIA Main / TVB-009 Transition Period
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/165 | 0/148 | 0/72 | 0/71
Serious Adverse Events (participants affected / at risk) | 8/166 | 6/165 | 5/148 | 0/72 | 1/71
Other Adverse Events (participants affected / at risk) | 123/166 | 108/165 | 42/148 | 20/72 | 11/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TVB-009 Main Treatment Period (N=166) | PROLIA Main Treatment Period (N=165) | TVB-009 Main / TVB-009 Transition Period (N=148) | PROLIA Main / PROLIA Transition Period (N=72) | PROLIA Main / TVB-009 Transition Period (N=71)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective periostitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TVB-009 Main Treatment Period (N=166) | PROLIA Main Treatment Period (N=165) | TVB-009 Main / TVB-009 Transition Period (N=148) | PROLIA Main / PROLIA Transition Period (N=72) | PROLIA Main / TVB-009 Transition Period (N=71)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 5 (5) | 2 (2) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 17 (17) | 22 (22) | 3 (3) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 7 (7) | 9 (9) | 4 (4) | 5 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (6) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Vitamin D decreased (Investigations) | 10 (10) | 5 (5) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 14 (14) | 19 (19) | 4 (4) | 2 (2) | 2 (2)
Vitamin D deficiency (Metabolism and nutrition disorders) | 34 (34) | 21 (21) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (14) | 13 (13) | 4 (4) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 6 (6) | 8 (8) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (10) | 3 (3) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 16 (16) | 15 (15) | 4 (4) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 8 (8) | 8 (8) | 1 (1) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must receive sponsor approval for all publications of study results.

DOCUMENTS (2):
  • Study Protocol (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT04729621/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/21/NCT04729621/SAP_001.pdf